CLINICAL TRIAL: NCT01988311
Title: Pilot Study: Effects of Psilocybin on Behavior, Psychology and Brain Function in Long-term Meditators
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Roland Griffiths, Professor, Johns Hopkins University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NA_00047665
Record Dates: First submitted 2013-10-18; First posted 2013-11-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Psilocybin; Hallucinogens; Pharmacologic Actions; Central Nervous System Agents; Therapeutic Uses; Psychotropic Drugs
Keywords: Psilocybin; Hallucinogens; Pharmacologic Actions; Central Nervous System Agents; Therapeutic Uses; Psychotropic Drugs
MeSH Terms: interventions — Psilocybin

ARMS (3):
- Drug Only (Experimental): psilocybin dose manipulation as described in the protocol
  Interventions: Drug: psilocybin
- Cognitive/Behavioral Tasks Only (No Intervention)
- Imaging Only (No Intervention)

INTERVENTIONS:
Drug: psilocybin — dose manipulation as described in the protocol
  Arms: Drug Only

SUMMARY:
This is a pilot study to finalize methods for a larger study being planned for the future. This research is being done to characterize performance of tasks, brain functioning, and the effects of psilocybin in individuals with a long-term meditation practice.

There are three different parts of the pilot study:

1. Effects of psilocybin on psychological function: This version of the pilot study will involve 1 or 2 day-long psilocybin sessions, and several meetings and data assessment visits. You will make a total of about 5 to 10 visits to our research unit (the BPRU on the Johns Hopkins Bayview Campus).
2. Performance on behavioral and cognitive tasks: This version of the pilot study will involve completing various behavioral and cognitive tasks at our research unit. You will make a total of about 1-10 visits to our research unit (the BPRU on the Johns Hopkins Bayview Campus).
3. Brain functioning: This version of the study will involve 1 to 3 brain imaging (MRI) measurements. You will make a total of about 2 to 5 visits to our research unit (the BPRU on the Johns Hopkins Bayview Campus). The MRI measurements will be taken at the F.M. Kirby Research Center at the Kennedy Krieger Institute (across the street from the Johns Hopkins Hospital).

People who are between the ages of 25 and 80 years old, who have a current, regular meditation practice, and who meet the medical requirements may join.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 80 years old
* Have given written informed consent
* Have some college-level education (college degree preferred)
* Be healthy and psychologically stable as determined by screening for medical and psychiatric problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on session days.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, within 24 hours of each drug administration. The exception is caffeine. Participants will be required to be non-smokers.
* Agree not to take any PRN medications on the mornings of drug sessions
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.

Exclusion Criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), or TIA in the past year
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting pharmacological effect on serotonin neurons or medications that are MAO inhibitors. For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* More than 20% outside the upper or lower range of ideal body weight according to Metropolitan Life height and weight table

Psychiatric Exclusion Criteria:

* Current or past history of meeting DSM-IV criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I or II Disorder
* Current or past history within the last 5 years of meeting DSM-IV criteria for alcohol or drug dependence (excluding caffeine and nicotine) or severe major depression
* Have a first or second-degree relative with Schizophrenia, Psychotic Disorder (unless substance induced or due to a medical condition), or Bipolar I or II Disorder
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin

fMRI Exclusion Criteria:

* Head trauma
* Claustrophobia
* Cardiac pacemaker
* Implanted cardiac defibrillator
* Aneurysm brain clip
* Inner ear implant
* Artificial heart valve (last 6 weeks)
* Prior history as a metal worker and/or certain metallic objects in the body

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Persisting Effects Questionnaire | 8 weeks post session
  Measures changes in spirituality, personal well-being, relationships, and emotions.
Hood Mysticism Scale | End of session day
  Measures subjective experience associated with classical mystical experiences.
States of Consciousness Questionnaire | End of session day
  Measures subjective experience associated with classical mystical experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] DiRenzo D, Barrett FS, Perin J, Darrah E, Christopher-Stine L, Griffiths RR. Impact of Psilocybin on Peripheral Cytokine Production. Psychedelic Med (New Rochelle). 2024 Jun 17;2(2):109-115. doi: 10.1089/psymed.2023.0039. eCollection 2024 Jun. PMID 40051582